CLINICAL TRIAL: NCT00050401
Title: Impact of Aggressive Empiric Antibiotic Therapy on the Emergence of Antimicrobial Resistance During the Treatment of Ventilator-associated Pneumonia
Brief Title: Ventilator-Associated Pneumonia/Hospital-Acquired Pneumonia Requiring Mechanical Ventilatory Support
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3591IL/0082
Record Dates: First submitted 2002-12-08; First posted 2002-12-10 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Pneumonia
Keywords: ventilator-associated; nosocomial
MeSH Terms: conditions — Pneumonia | interventions — Meropenem

INTERVENTIONS:
Drug: MERREM I.V. 2g as a 3 hour infusion every 8 hours
Drug: vancomycin I.V. 1 g every 12 hours
Drug: tobramycin I.V. 5 mg/kg every 24 hours
Drug: MERREM I.V. 1g as a 30 minute infusion every 8 hours
Drug: MERREM I.V. 500 mg as a 3 hour infusion every 8 hours

SUMMARY:
The purpose of the study is to find out if high dose antibiotic (meropenem, MERREM® I.V.), along with another drug called an aminoglycoside (a different type of antibiotic) is effective in decreasing or reducing the rate of antibiotic resistant Pseudomonas aeruginosa, Acinetobacter (germs that can cause pneumonia), and the rate of resistance in other difficult to treat germs which may cause hospital-acquired pneumonia requiring mechanical ventilatory support. The study hopes to show that by increasing the amount of meropenem administered and increasing the duration of infusion (release of the drug into the bloodstream), levels of the drug will stay at target levels in the bloodstream and decrease the ability of difficult to treat germs to resist, or not be killed by, the treatment using this antibiotic (meropenem) or other antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Onset or exacerbation of pneumonia at least 72 hours after admission to an acute care facility or onset of pneumonia in a nursing home or rehabilitation facility with subsequent transfer to an acute care facility
* Diagnosis of hospital-acquired pneumonia requiring mechanical ventilatory support
* Patient or Patient's legal guardian must sign written informed consent for study participation, pretreatment, and Day 7 bronchoscopy

Exclusion Criteria:

* Patients with hospital-acquired pneumonia caused by pathogens resistant to MERREM
* Patients with allergies to cephalosporins, penicillins and carbapenems
* Patients taking anticonvulsant therapy for a known seizure disorder
* Patients with lung cancer
* Patients with cystic fibrosis, acquired immune deficiency syndrome (AIDS), neutropenia, active tuberculosis, or patients taking immunosuppressive therapy in preparation for or following an organ transplant.
* Patients who are pregnant or breast feeding
* Patients who are unlikely to survive
* Patients with certain infections in another area requiring treatment with additional antibiotics
* Patients with other underlying conditions that would make it difficult to interpret response to study drug.
* Patients who have been part of another clinical study 30 days before entry into this study.
* Patients with hypotension (systolic BP < 85mmHg) or acidosis (arterial pH <7.25 or serum bicarbonate <15 mg/dl) despite attempts at fluid resuscitation
* Patients with profound hypoxia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2002-07; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Phoenix, Arizona
  - Newark, Delaware
  - Indianapolis, Indiana
  - Boston, Massachusetts
  - Lebanon, New Hampshire
  - Albany, New York
  - New York, New York
  - Stony Brook, New York
  - Cincinnati, Ohio
  - San Antonio, Texas